CLINICAL TRIAL: NCT03119727
Title: Clinical Evaluation of the Automatic Oxygen Adjustment by FreeO2 in a Medical Population in Hospital
Brief Title: Clinical Evaluation of FreeO2 (Version 4) in All Patients Receiving Oxygen
Acronym: FreeO24G
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, François Lellouche, Principal Investigator, Laval University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21342
Record Dates: First submitted 2017-04-12; First posted 2017-04-19 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Respiratory Disease; Respiratory Failure; COPD Exacerbation; Asthma; Pneumonia
MeSH Terms: conditions — Respiration Disorders; Respiratory Insufficiency; Asthma; Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Automated oxygen adjustment (Other): All patient in this study have automatic oxygen titration and automatic oxygen weanning
  Interventions: Device: FreeO2

INTERVENTIONS:
Device: FreeO2 — All include patients will have automatic administration of oxygen by FreeO2 up to 3 day or until weaning of oxygen adminisatrion

SUMMARY:
Evaluation of automatic titration of oxygen with a new version of FreeO2 (V4)

DETAILED DESCRIPTION:
In the previous studies, the investigators used many times automatic titration of oxygen on spontanous breathing patient (FreeO2 device) with a prototype develop in our lab in collaboration with Laval university. In this study, we want to evaluate the new version of the FreeO2 device (V4)

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years old
* Patient receiving oxygen between 1 to 6 lpm for medical pathology
* Admitted to a medical service for less than 72 hours (emergency room not included)

Exclusion Criteria:

* Unreliable SpO2 signal
* Emergency or intensive care hospitalization
* Absence of NIV or intubation criteria at baseline
* Sleep apnea not paired
* Long-term Oxygen Therapy
* Active delirium and cognitive impairment preventing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2020-11-06 (Actual)

PRIMARY OUTCOMES:
% of time in the set SpO2 target | During 3 days of hospitalization or until Oxygen weaning
  Continuous SpO2 monitoring (1 data each second) will be recorded, the % of time within the SpO2 target±2% set by the physician will be considered (Time in the target±2/Total recording time)

SECONDARY OUTCOMES:
Oxygenation data | 3 hospitalisations day or until Oxygen weaning
  the % of time with hyperoxia (SpO2 > SpO2 target+5%), the % of time with severe hypoxemia (SpO2 <85%) the % of time without SpO2 signal, the % of time with oscillations of SpO2 values, comparison of Wired SpO2 vs Bluetooth SpO2, Daily variations of oxygen flows J1, J2 and J3
  % Weaning> 50% relative baseline,% complete weaning of O2

CONTACTS AND LOCATIONS:
Locations (1):
- IUCPQ-UL, Québec, Quebec, Canada